CLINICAL TRIAL: NCT02943525
Title: Vaginal Packing After Laparoscopic Sacrocolpopexy; Patient Pain and Satisfaction in Short Follow-up and Surgery Outcome and Complications in One Year Follow-up
Brief Title: Vaginal Packing After Laparoscopic Sacrocolpopexy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Zdenek Rusavy, M.D., Ph.D., Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PACKING
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Vaginal Packing Following Laparoscopic Sacrocolpopexy; Pelvic Organ Prolapse
Keywords: vaginal packing; pelvic organ prolapse; pain and satisfaction
MeSH Terms: conditions — Pelvic Organ Prolapse; Pain; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- packing (Experimental): Patients after laparoscopic sacrocolpopexy with a vaginal packing at the end of surgery
  Interventions: Procedure: vaginal packing
- no packing (No Intervention): Patients after laparoscopic sacrocolpopexy without a vaginal packing at the end of surgery

INTERVENTIONS:
Procedure: vaginal packing — Packing vagina with a Boric acid soaked gauze at the end of surgery
  Arms: packing

SUMMARY:
Vaginal packing is used routinely following vaginal reconstructive surgery, however, no recommendation regarding vaginal packing after laparoscopic sacrocolpopexy exists. Despite little data to support the practice, purported benefits better positioning and fixation of the mesh, improving incorporation of the mesh by its fixation and reduced blood loss. Patients often complain of discomfort associated with the packing or its removal. The aim of this randomized controlled is to compare the subjective impressions of pain and bother in women undergoing laparoscopic sacrocolpopexy treated with and without packing. The investigators also aim to assess differences in postoperative bacteriuria, urine retention and hemoglobin levels on day 5 after the surgery and surgery outcome and complications at one year after the surgery in those with and without packing.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic sacrocolpopexy without a suburethral sling
* Pelvic organ prolapse stage > 2
* Speak and read Czech
* Can to understand the informed consent

Exclusion Criteria:

* Any other surgery than sacrocolpopexy
* Concurrent hysterectomy or opening of the vagina during the surgery.
* Vaginal, uterine, cervical or ovarian malignancy
* Clotting disorder, taking anticoagulation
* Having intraoperative blood loss greater than 500 ml

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain assessed using VAS | The first post-operative day before extraction of the packing
  Visual analog scale (VAS)
Satisfaction with the overall postoperative course assessed using VAS | Postoperative day 5
  VAS
Prolapse recurrence | 1 year after the surgery
  Pelvic Organ Prolapse Quantification System (POP-Q) classification - the most descending compartment >-1cm from hymen
Surgery related complications | From the surgery until 1 year after the surgery
  According to the International Continence Society / International UroGynecology Association Joint Terminology and Classification Report of the complications related directly to the insertion of prostheses (meshes, implants, tapes) & grafts in female pelvic floor surgery
Postoperative pain assessed using the McGill Questionnaire | The first post-operative day before extraction of the packing
  McGill Questionnaire

SECONDARY OUTCOMES:
Number of analgesics used | From the end of the surgery until the first postoperative day
Positive urine culture | Postoperative day 5
Satisfaction with surgery assessed using VAS | Postoperative day 1 before packing extraction
  VAS

CONTACTS AND LOCATIONS:
Overall Officials: Zdenek Rusavy, MD PhD, Principal Investigator — Medical Faculty in Pilsen, Charles University
Locations (1):
- Department of Obstetrics and Gynecology, Charles University Hospital, Pilsen, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thiagamoorthy G, Khalil A, Cardozo L, Srikrishna S, Leslie G, Robinson D. The value of vaginal packing in pelvic floor surgery: a randomised double-blind study. Int Urogynecol J. 2014 May;25(5):585-91. doi: 10.1007/s00192-013-2264-y. Epub 2013 Dec 6. PMID 24310987
- [Background] Westermann LB, Crisp CC, Oakley SH, Mazloomdoost D, Kleeman SD, Benbouajili JM, Ghodsi V, Pauls RN. To Pack or Not to Pack? A Randomized Trial of Vaginal Packing After Vaginal Reconstructive Surgery. Female Pelvic Med Reconstr Surg. 2016 Mar-Apr;22(2):111-7. doi: 10.1097/SPV.0000000000000238. PMID 26825408
- [Derived] Rusavy Z, Marinic Veverkova A, Smazinka M, Kalis V. Vaginal packing after laparoscopic sacrocolpopexy - postoperative pain and satisfaction: a randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2026 Jan;316:114815. doi: 10.1016/j.ejogrb.2025.114815. Epub 2025 Nov 5. PMID 41202691
- [Derived] Rusavy Z, Marinic Veverkova A, Smazinka M, Kalis V. Vaginal packing after laparoscopic sacrocolpopexy and surgical outcome after one year: A randomized controlled trial. Acta Obstet Gynecol Scand. 2025 Dec;104(12):2331-2338. doi: 10.1111/aogs.70067. Epub 2025 Oct 10. PMID 41070594